CLINICAL TRIAL: NCT01110629
Title: Randomized, Double-blind, Parallel-group, Placebo-controlled Study of Lanthanum Carbonate 750 to 2250 mg in Patients With Chronic Kidney Disease Not on Dialysis Who Develop Hyperphosphatemia
Brief Title: Study in Chronic Kidney Disease (CKD) Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14817
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Hyperphosphatemia
Keywords: Chronic kidney disease not on dialysis; Lanthanum carbonate
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Fosrenol (Lanthanum Carbonate, BAY77-1931)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosrenol (Lanthanum Carbonate, BAY77-1931) — Daily dose: 750-2250mg 3 times a dayfor 8 weeks.
  Arms: Arm 1
Drug: Placebo — daily dose: 3 tablets TID for 8 weeks.
  Arms: Arm 2

SUMMARY:
The objective of this study is to investigate the efficacy and safety of lanthanum carbonate 750 to 2,250 mg in Japanese Chronic Kidney Disease Stage 3, 4 and 5 subjects not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 years or above at the time of informed consent
* Chronic Kidney Disease patients with Epidermal growth factor receptor (eGFR) under 60 ml/min/1.73m2 (stage 3, 4 and 5) who have not been on dialysis
* Patients who had been in the care of a physician for Chronic Kidney Disease for >2 months and was not expected to begin dialysis for at least 4 months
* Patients with serum phosphate levels 5.6 mg/dL to 11.0 mg/dL at Week -4 (Visit 1) or Week -2 (Visit 2)

Exclusion Criteria:

* Patients with hypocalcemia or hypercalcemia (corrected serum calcium level of < 7.0 mg/dL or >/- 11.0 mg/dL) at Week -2 (Visit 2).
* Significant renal impairments
* Had acute renal failure within 3 months of Run-in period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The change from baseline in serum phosphate concentrations | Week 8

SECONDARY OUTCOMES:
Achievement of target serum phosphate level (2.7 to 4.6 mg/dL) | Week 0, Week 2, Week 4, Week 6, Week 8
Change in serum Calcium x Phosphor product | Week 0, Week 2, Week 4, Week 6, Week 8
Serum intact PTH level | Week 0, Week 2, Week 4, Week 6, Week 8
Phosphate excretion in urine | Week 0, Week 4, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (31):
- Japan (31):
  - Anjo, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Toyohashi, Aichi-ken
  - Yatomi, Aichi-ken
  - Kamogawa, Chiba
  - Kisarazu, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Kyoto, Kyoto
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Sakai, Osaka
  - Saga, Saga-ken
  - Shizuoka, Shizuoka
  - Tokushima, Tokushima
  - Koto, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Shinagawa, Tokyo
  - Wakayama, Wakayama

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Takahara Y, Matsuda Y, Takahashi S, Shigematsu T; Lanthanum Carbonate Study Group. Efficacy and safety of lanthanum carbonate in pre-dialysis CKD patients with hyperphosphatemia: a randomized trial. Clin Nephrol. 2014 Sep;82(3):181-90. doi: 10.5414/cn108269. PMID 25079863